CLINICAL TRIAL: NCT04105205
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Apramycin Administered Intravenously in Healthy Adults.
Brief Title: First-In-Human Study of Apramycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juvabis AG (Industry)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: JUV18-01
Record Dates: First submitted 2019-09-12; First posted 2019-09-26 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers
Keywords: Anti-Bacterial Agents
MeSH Terms: interventions — apramycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apramycin injection in escalating doses (Experimental): Apramycin, solution for infusion.
  Interventions: Drug: Apramycin injection
- Placebo (Placebo Comparator): Physiological saline, solution for infusion.
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Apramycin injection — 30-min infusion
  Arms: Apramycin injection in escalating doses
Drug: Placebo injection — 30-min infusion
  Arms: Placebo

SUMMARY:
This is a first-in-human study to assess the safety, tolerability and pharmacokinetics of escalating single doses of apramycin. This trial will be conducted as a single ascending dose trial in up to 5 sequential dose cohorts (group-comparison). Each cohort will consist of 8 healthy subjects, 6 will receive apramycin and 2 placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects of non-childbearing potential, 18-45 years of age (both inclusive), body mass index 18.0 - 29.9 kg/m2 (inclusive) and body weight from 50 to 100 kg (inclusive).
* Glomerular filtration rate (GFR) ≥ 90 mL/min /1.73 m2.
* Subjects with systemic hearing, with air conduction thresholds no worse than 20 decibels (dB) hearing loss for the frequencies 0.5-1-2-4-6-8 kilohertz (kHz) bilaterally and, no threshold asymmetry ≥ 20 dB at any frequency, normal (reproducibility 70% or better) transient evoked otoacoustic emissions (TEOAE).
* From the signing of the informed consent until the last follow-up visit, subjects must be willing to avoid exposure to loud noise and Subjects must be willing to avoid excessive physical exercise within 48 h prior to dosing.
* Normal blood pressure and pulse rate, ECG recording without clinically significant abnormalities.
* Thyroid-stimulating hormone, free triiodothyronine and free thyroxine within the reference ranges.
* Having had no febrile or infectious illness for at least 7 days prior to the first administration of the Investigational medicinal product (IMP) of the study.
* Normal microscopic findings in the ears, normal tympanic membrane mobility and stapedial reflex present.

Exclusion Criteria:

* Vegetarian or vegan.
* Demonstrating excess in xanthine consumption.
* More than low-risk alcohol consumption (men: ≥24 g of pure alcohol regularly per day; women: ≥12 g of pure alcohol regularly per day).
* Any history of alcohol or drug abuse or a positive urine drug screen test. Positive alcohol breath test.
* Consumption of xanthine-containing food or beverages within 48 h before dosing.
* Smokers smoking more than 10 cigarettes or equivalent per day.
* Exposure to loud noise within 3 days prior to drug administration.
* Taking any medication on a regular basis, with the exception of solitary doses of up to 1000 mg paracetamol.
* Use of any investigational drug product within 30 days or 5 half-lives before screening.
* Use of aminoglycosides or other antibiotics within 3 months prior to screening.
* Use of neuromuscular blocking agents within 1 week or 5 half-lives prior to screening.
* Use of potentially nephrotoxic medication 2 weeks prior to the drug administration.
* Any history of drug hypersensitivity, asthma, urticaria or other severe allergic diathesis as well as hay fever with ongoing symptoms.
* Any history of hypersensitivity to aminoglycosides.
* Any history or signs of acute, chronic or recurrent metabolic, renal, hepatic, pulmonary, gastrointestinal, neurological, neuromuscular disorders, endocrinological, immunological, psychiatric or cardiovascular disease, myopathies, and bleeding tendency.
* Problems with hearing and/or balance.
* Previous injury or surgery to the middle or inner ears, family history of hearing loss before the age of 60.
* Genetic predisposition to aminoglycoside-driven ototoxicity.
* Laboratory values outside the reference range that are of clinical relevance.
* Positive test for HIV antibodies, hepatitis B-virus surface antigen, or anti-hepatitis C-virus antibodies.
* Blood or plasma donation of 500 mL within 3 months or more than 100 mL within 30 days before signing an informed consent to this trial.
* Judged by the investigator to have occupational noise exposure of high risk during the trial.
* Positive test for SARS-CoV-2.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Type and incidence of treatment-emergent adverse events (TEAEs) until 2 weeks after dosing. | until 2 weeks after dosing
Type and incidence of TEAEs related to auditory and vestibular function tests. | until 3 months after dosing
Number of subjects with clinically significant vital sign measurement blood pressure. | until 2 weeks after dosing
  Frequency is defined as number of subjects with clinically significant observations.
Number of subjects with clinically significant vital sign measurement pulse rate. | until 2 weeks after dosing
  Frequency is defined as number of subjects with clinically significant observations.
Number of subjects with clinically significant observation in physical examination. | until 2 weeks after dosing
  Frequency is defined as number of subjects with clinically significant observations.
Number of subjects with clinically significant changes in clinical laboratory parameters. | until 2 weeks after dosing
  Frequency is defined as number of subjects with clinically significant observations.
Number of subjects with clinically significant changes in ECG parameters. | until 2 weeks after dosing
  ECG parameters include heart rate and PQ, QT, RS. Frequency is defined as number of subjects with clinically significant observations.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Schultz, Dr.med., Principal Investigator — CRS Clinical Research Services Mannheim GmbH
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roch M, Sierra R, Sands K, Martins WMBS, Schrenzel J, Walsh TR, Gales AC, Andrey DO. Vertical and horizontal dissemination of an IncC plasmid harbouring rmtB 16S rRNA methylase gene, conferring resistance to plazomicin, among invasive ST258 and ST16 KPC-producing Klebsiella pneumoniae. J Glob Antimicrob Resist. 2021 Mar;24:183-189. doi: 10.1016/j.jgar.2020.12.006. Epub 2020 Dec 26. PMID 33373732